CLINICAL TRIAL: NCT03378583
Title: Is Ultrasound-guided Left Paratracheal Esophagus Pressure More Effective Than Cricoid Pressure to Prevent Gastric Insufflation During Positive Pressure Ventilation ?
Brief Title: Prevention of Gastric Insufflation During Positive Pressure Ventilation ?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Chair of department of anesthesia and intensive care medicine, University of Liege
Other Study IDs: ULGANESGAU001
Record Dates: First submitted 2017-12-14; First posted 2017-12-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Complication of Ventilation Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control,: control normal ventilation
- sellick,: ventilation while sellick manoeuvre is applied
- low paratracheal esophagus compression: ventilation while low paratracheal esophagus compression is applied

SUMMARY:
Evaluation of a new method to prevent gastric insufflation

DETAILED DESCRIPTION:
After Ethics Committee approval of the University of Liège and written informed consent, 90 ASA 1-2 patients aged 18-65 years and scheduled for elective surgery under general anesthesia will be enrolled in the study. Exclusion criteria are body mass index (BMI) above 35; meeting criteria for difficult ventilation and/or intubation, such as oropharyngeal pathology or facial or cervical abnormalities; and risk for aspiration or previous gastric surgery. Patients will be randomly allocated 1:1:1 (30 patients/group) by the method of sealed envelopes to left low paratracheal esophageal compression (LPEC), cricoid pressure (CP), or no pressure intervention (Control). Neck circumference will be measured. No premedication will be given prior to the study interventions.

Part 1: Ultrasound assessment of the esophagus at the left lower paratracheal level

Esophageal examinations will be conducted by ultrasound with the patient supine and head in neutral position. Feasibility of imaging and compressing the esophagus approximately 2-3 cm above the clavicle was assessed as follows:

A linear ultrasound probe (Applio XG iStyle Toshiba with a 14-7 Mhz) was positioned in a transverse (axial) orientation over the left paratracheal area (Figure 1(A)), 2-3 cm above the clavicle. The position of the esophagus in relation to the trachea (left, right or not seen) will be recorded. Once the esophagus will be identified, the antero-posterior diameter (mm) will be measured and compared before and after applying an estimated pressure of 30 N (as described below) or until a bony contact will be established with the transducer. Esophageal compression will be re-assessed using a paramedian sagittal plane between the trachea and the sternocleidomastoid muscle with the esophagus in sagittal plane. The antero-posterior diameter (mm) measurements will be repeated before and after applying pressure with the transducer. Three consecutive measures for each probe position were recorded.

Part 2: Assessment of the presence of gastric (antral) air With the patients in supine position, a curvilinear transducer (Applio XG iStyle Toshiba with an 8-5 MHz) will be placed on the epigastrium in a paramedian sagittal orientation to identify the antrum. 9 The cross-sectional area of the antrum was measured at the level where both the aorta and upper mesenteric artery were visible. Three consecutive measures were taken (a) before the induction of anesthesia and (b) after 3 min of PPV via face mask. The presence of gastric air insufflation is defined as an increase in cross-sectional area and/or presence of artifacts in the antrum (comet tail, posterior acoustic shadow). 9 These assessments will be performed by a sonographer, blinded to group allocation by a surgical drape placed between the thorax and the abdomen.

Pressure maneuvers Two anesthesiology residents, not informed of the study outcome measurements, will be trained to apply sustained pressure of 30 ± 5 N using an electronic dynamometer (MicroFET2; Hoogan Industries, West Jordan, Utah), until 10 consecutive maneuvers will be measured successfully (30 ± 5 N). For cricoid pressure, the cartilage will be compressed with the thumb and index fingers toward the vertebral bodies (Sellick). For LPEC, the thumb will be placed over the base of the neck on the left side of the trachea 2-3 cm above the clavicle and medial to the sternocleidomastoid muscle (Figure 1(B)).

ASA monitoring will be applied, and anesthesia will be induced with propofol 2.5 mg/kg administered over 45 sec. Remifentanil will be administered with an infusion pump (2 to 3 μg/kg over 60 sec during induction, followed by continuous infusion of 0.05μg /kg/min). After general anesthesia will be induced, PPV was accomplished with a face-mask in pressure-control mode while maintaining a positive inspiratory pressure of 25 cm H2O, (Zeus ventilator, Dräger, Lübeck, Germany). The ventilator settings will be 100% oxygen, I:E ratio 1:2, 15 breaths/min, no positive end-expiratory pressure. Adequacy of ventilation will be documented by chest raise and capnography. Antral measurements will be taken after 3 min of face-mask ventilation by a sonographer blinded to group assignment. Thereafter, the management of anesthesia care will be continued as per institutional standards.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery under general anesthesia

Exclusion Criteria:

* body mass index above 35 meeting criteria for difficult ventilation and /or intubation risk for aspiration or gastric surgery

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients undergoing anesthesia under general anesthesia
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2017-03-22 (Actual); Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
gastric volume | within 10 min of induction of anesthesia
  With the patients in supine position, a curvilinear transducer (Applio XG iStyle Toshiba with an 8-5 MHz) will be placed on the epigastrium in a paramedian sagittal orientation to identify the antrum. The cross-sectional area of the antrum will be measured at the level where both the aorta and upper mesenteric artery will be visible

SECONDARY OUTCOMES:
diameter of the esophagus | within 10 min of induction of anesthesia
  A linear ultrasound probe (Applio XG iStyle Toshiba with a 14-7 Mhz) will be positioned in a transverse (axial) orientation over the left paratracheal area (Figure 1(A)), 2-3 cm above the clavicle. The position of the esophagus in relation to the trachea (left, right or not seen) will be recorded. When the esophagus will be identified, the antero-posterior diameter (mm) will be measured and compared before and after applying an estimated pressure of 30 N.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Liege, Liège, Liege, Belgium

IPD SHARING:
Plan to Share IPD: No